CLINICAL TRIAL: NCT00295958
Title: Phase II Evaluation of Peptide Immunization and LMB-2 in Metastatic Melanoma
Brief Title: LMB-2 Immunotoxin and Vaccine Therapy in Treating Patients With Metastatic Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Masking: None | Purpose: Treatment
Other Study IDs: 060041; 06-C-0041; NCI-7542; NCI-P6702; CDR0000462165; NCT00263510 (obsolete NCT alias)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma (Skin); Non-melanomatous Skin Cancer
Keywords: recurrent melanoma; stage IV melanoma; skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin; MART-1 Antigen; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: LMB-2 immunotoxin
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: The LMB-2 immunotoxin can find tumor cells and kill them without harming normal cells. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving LMB-2 immunotoxin together with vaccine therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving LMB-2 immunotoxin together with vaccine therapy works in treating patients with metastatic melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine objective clinical response in patients with progressive, unresectable metastatic melanoma treated with recombinant LMB-2 immunotoxin and peptide vaccination comprising gp100:209-217 (210M) antigen, MART-1:27-35 antigen, and Montanide ISA-51.

Secondary

* Determine changes in levels of CD4+, CD25+ regulatory T cells in peripheral blood before and after treatment in patients treated with this regimen.
* Determine the ability of recombinant immunotoxin LMB-2 to augment peptide vaccination in these patients.
* Determine the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive LMB-2 immunotoxin IV over 30 minutes twice on days 1-3. Patients then receive peptide vaccinations comprising gp100:209-217 (210M) antigen emulsified in Montanide ISA-51 subcutaneously (SC), and MART-1:27-35 vaccine emulsified in Montanide ISA-51 SC on days 4, 5, 6, and 24-27 (course 1). After week 8, patients achieving tumor response may receive 1 additional course in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically in the absence of disease progression.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma

  * Unresectable disease
  * Progressive disease while receiving standard therapy (e.g., interleukin-2 or dacarbazine)
* HLA-A0201 positive
* Measurable disease
* The following are not allowed:

  * Resectable local/regional disease
  * Patients whose serum neutralizes LMB-2 in tissue culture, due either to antitoxin or antimouse-immunoglobulin G antibodies (> 75% of the activity of 1 ug/mL of LMB-2)
  * Received LMB-2 on another trial

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy more than 3 months
* WBC ≥ 3,000/mm^3
* Absolute lymphocyte count > 500/mm^3
* Platelet count ≥ 90,000/mm^3
* Bilirubin ≤ 2.0 mg/dL (≤ 3.0 mg/dL for patients with Gilbert's syndrome)
* AST and ALT ≤ 2.5 times normal
* Albumin ≥ 3.0 g/dL
* No hepatitis B surface antigen or hepatitis C positivity
* Creatinine ≤ 1.4 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* Ejection fraction ≥ 45% by echocardiogram or thallium stress test (for patients > 50 years of age OR who have a history of cardiovascular disease)
* LVEF ≥ 45%
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No known HIV positivity
* No autoimmune disease
* No immunodeficiency
* No other malignancies
* Must be willing to undergo leukapheresis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 12 weeks since prior monoclonal antibody therapy
* More than 3 weeks since prior and no concurrent systemic therapy for cancer
* No concurrent chronic anticoagulant therapy
* No concurrent systemic steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-12; Primary Completion 2006-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Objective clinical response rate

SECONDARY OUTCOMES:
Changes in levels of CD4+, CD25+ regulatory T cells
Ability of LMB-2 to augment peptide vaccination
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland